CLINICAL TRIAL: NCT05801510
Title: Cognitive Muscular Therapy for People Awaiting Knee Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Stephen Preece, Professor of Biomechanics and Rehabilitation, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMT-TKR-317409
Record Dates: First submitted 2023-03-17; First posted 2023-04-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Cognitive Muscular Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: All partiticipants will receive seven sessions of CMT over a 7 week period. All participants will complete questionnaires at baseline and at 10 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The treatment group will receive seven sessions of CMT over a 14 week period.
  Interventions: Behavioral: Cognitive Muscular Therapy for knee pain

INTERVENTIONS:
Behavioral: Cognitive Muscular Therapy for knee pain — Psychologically informed physiotherapy which uses biofeedback training to reduce muscle overactivity and improve postural control and also encourages people to change the way they react to pain.

SUMMARY:
The primary aim will seek to understand whether Cognitive Muscular Therapy (CMT) could provide pain relief for people on a waiting list for joint replacement.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a chronic long-term condition that results in pain, disability and reduced quality of life. While current guidelines focus on the use of exercises to improve strength, there is clear evidence that people with knee osteoarthritis over-activate their muscles during functional tasks. Through NIHR funding the investigators have developed a new behavioural intervention for people with KOA- Cognitive Muscular Therapy (CMT). CMT aims to reduce overactivity of the knee muscles and change the way people react to pain. Importantly, muscle overactivity has been linked to increased pain, elevated joint loading and a more rapid rate of cartilage loss. Our pilot data suggests CMT can reduce knee osteoarthritis pain. Specifically, the investigatorsobserved a 69% reduction in pain in 11 patients who received six sessions of CMT. The investigators have subsequently trained 5 NHS physiotherapists to deliver CMT and observed them deliver the intervention to 12 patients. These patients reported average improvements in pain of 85% after 7 sessions.The proposed project will seek to understand whether CMT could provide pain relief for people on a waiting list for joint replacement. The first stage of the project will seek to understand patient's and clinicians perceptions of knee osteoarthritis. This insight will allow us to map changes to CMT which will make it suitable for people on a waiting list for knee replacement. Following modification of the intervention, the investigators plan to recruit 24 participants from knee replacement waiting lists in Manchester, UK. All participants will recieve the CMT treatment and this will consist of seven sessions of CMT over a 7 week period. All participants will complete questionnaires at baseline and at 10 weeks and will be offered an interview to understand their experiences.

ELIGIBILITY:
Inclusion:

1. Above 40 years old
2. Speak and understand English sufficient to read the information sheet and sign the consent form
3. Ability to walk without any assistive device for at 20m (to ensure sufficient mobility to complete the intervention)
4. Radiological diagnosis of knee OA
5. On orthopaedic waiting but currently expected to wait at least 6 months for surgery (this will ensure that that the patient's care pathway is not affected)

Exclusion:

1. Dementia or other major cognitive impairment.
2. BMI >30 (as increased subcutaneous fat prevents collection of surface EMG signals)
3. Previous knee replacement
4. Any active systemic inflammatory disorders, such as rheumatoid arthritis with patient taking immunosuppressant drugs or steroids
5. Any balance disorders which may increase the risk of a fall
6. A history of rupture to the anterior cruciate ligament/ posterior cruciate ligament/ medial collateral ligament/ lateral collateral ligament
7. A diagnosis of psoriatic arthritis
8. A diagnosis of post traumatic arthritis for example after a previous tibial plateau/ patella fracture
9. A diagnosis of septic arthritis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain. | Change from Baseline to 10 weeks
  The extent of pain in the involved knee during five activities. Score 0-20 (0=no pain, 20=maximum pain)

SECONDARY OUTCOMES:
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) (full score) | Change from Baseline to 10 weeks
  To assess pain and function in the involved knee. Score 0-96 (0=no pain/full function, 96=maximum pain/lowest function)

OTHER OUTCOMES:
Change in Pain catastrophizing scale | Change from Baseline to 10 weeks
  Used to capture pain catastrophizing behaviours. Score 0-52 (0=no pain catastrophizing, 52=maximum pain catastrophizing)
Change in the EQ-5D-5L | Change from Baseline to 10 weeks
  Captures the patient's self-rated health. Score 0-1 ( 0= death,1= perfect health)
Change in the Health resource utilisation - custom questionnaire | Change from Baseline to 10 weeks
  To capture to use of health(care) resources
Change in the Oxford Knee Score | Change from Baseline to 10 weeks
  The Oxford Knee Score (OKS) is a 12-item patient-reported PRO specifically designed and developed to assess function and pain. Score- (0= severe arthritis, 60=satisfactory joint function
Change in the UCLA Activity Score | Change from Baseline to 10 weeks
  Used to capture activity levels. Score (1= low activity, 10= high activity)
Change in the Arthritis Self Efficacy Scale (ASES) | Change from Baseline to 10 weeks
  Capture self-efficacy in people with arthritis. Score (8= low self efficacy, 80= high self efficacy)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The investigtors may make the clinical data available through a document which will be linked to the final published journal paper

REFERENCES:
- [Background] Preece SJ, Brookes N, Williams AE, Jones RK, Starbuck C, Jones A, Walsh NE. A new integrated behavioural intervention for knee osteoarthritis: development and pilot study. BMC Musculoskelet Disord. 2021 Jun 8;22(1):526. doi: 10.1186/s12891-021-04389-0. PMID 34103040
- See also: Description of Cognitive Muscular Therapy — http://hub.salford.ac.uk/cognitive-muscular-therapy/